CLINICAL TRIAL: NCT00463242
Title: An 8-week, Multicenter, Randomized, Double-blind, Placebo- and Paroxetine-controlled Study of the Efficacy, Safety and Tolerability of Agomelatine 25 or 50 mg Given Once Daily in the Treatment of Major Depressive Disorder (MDD) Followed by a 52-week Open-label Treatment With Agomelatine 25 or 50 mg
Brief Title: A Placebo- and Paroxetine-controlled Study of the Efficacy, Safety and Tolerability of Agomelatine (25 or 50 mg) in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAGO178A2303
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
Keywords: agomelatine, Major Depressive Disorder, MDD, depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Agomelatine (Experimental): Dosing for each subject in this extension study began with the same dose (25 mg or 50 mg of agomelatine orally once daily) the subject was receiving at the end of Week 8, the week before this study began.
  Interventions: Drug: Agomelatine
- 2 (Active Comparator)
  Interventions: Drug: paroxetine
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Agomelatine — Either 25 mg or 50 mg agomelatine orally once daily
  Arms: Agomelatine
Drug: paroxetine
  Other Names: Paxil
  Arms: 2
Drug: placebo
  Arms: 3

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of agomelatine 25 mg or 50 mg per day and will compare agomelatine and paroxetine tolerability. Eligible patients will receive double-blind study medication for 8 weeks. One week after completion of the double-blind treatment phase there will be a single follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 through 70 years of age, inclusive
* Diagnosis of Major Depressive Disorder according to DSM-IV criteria
* HAM-D17 total score > or = 22 at Screening and Baseline

Exclusion Criteria:

* History of non-response to paroxetine
* Patients who have been previously treated with agomelatine
* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder, or obsessive compulsive disorder
* Any current Axis I disorder other than major depressive disorder which is the focus of treatment
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months
* Use of any psychoactive medication after the screening visit
* Female patients of childbearing potential who are not using effective contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 on the total score Hamilton Depression Rating Scale | 8 weeks

SECONDARY OUTCOMES:
To demonstrate less sexual dysfunction in patients with MDD receiving agomelatine compared to paroxetine, as measured by the change from baseline to Week 8 on the total score of the Arizona Sexual Experience Scale (ASEX). | 8 weeks
Proportion of patients who demonstrate clinical improvement where improvement is defined by a score of 1 or 2 on the Clinical Global Impression Improvement (CGI-I) scale at Week 8. | 8 weeks
Proportion of patients with MDD who achieve remission, | 8 weeks
Change from baseline to Week 8 on the total score and Anxiety subscale of the Hospital Anxiety and Depression Scale (HAD). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (43):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, National City, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Pico Rivera, California
  - Novartis Investigative Site, Redlands, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Joliet, Illinois
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Fall River, Massachusetts
  - Novartis Investigative Site, Okemos, Michigan
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Willingboro, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Corvallis, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Media, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Friendswood, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Herndon, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Bellevue, Washington
  - Novartis Investigative Site, Waukesha, Wisconsin
- Novartis Investigative Site, Hato Rey, Puerto Rico

REFERENCES:
- See also: Results for CAGO178A2303 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2659